CLINICAL TRIAL: NCT06447012
Title: Development of a Novel Real Time Computer Assisted Colonoscopy Diagnostic Tool for Colorectal Polyps: Lesion Diagnosis and Personalised Patient Management
Brief Title: Artificial Intelligence Development for Colorectal Polyp Diagnosis
Status: Recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 323988
Record Dates: First submitted 2024-05-07; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Polyp of Colon; Colorectal Polyp
Keywords: Artificial Intelligence; Computer assisted diagnosis (CADx); Colorectal cancer; Colorectal polyp; Machine learning
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Colonoscopy — No intervention required from this study, however images will be obtained from patient presenting for colonoscopy

SUMMARY:
Accurate classification of growths in the large bowel (polyps) identified during colonoscopy is imperative to inform the risk of colorectal cancer. Reliable identification of the cancer risk of individual polyps helps determine the best treatment option for the detected polyp and determine the appropriate interval requirements for future colonoscopy to check the site of removal and for further polyps elsewhere in the bowel.

Current advanced endoscopic imaging techniques require specialist skills and expertise with an associated long learning curve and increased procedure time. It is for these reasons that despite being introduced in clinical practice, uptake of such techniques is limited and current methods of polyp risk stratification during colonoscopy without Artificial intelligence (AI) is suboptimal. Approximately 25% of bowel polyps that are removed by major surgery are analysed and later proved to be non-cancerous polyps that could have been removed via endoscopy thus avoiding anatomy altering surgery and the associated risks. With accurate polyp diagnosis and risk stratification in real time with AI, such polyps could have been removed non-surgically (endoscopically). Current Computer Assisted Diagnosis (CADx, a form of AI) platforms only differentiate between cancerous and non cancerous polyps which is of limited value in providing a personalised patient risk for colorectal cancer. The development of a multi-class algorithm is of greater complexity than a binary classification and requires larger training and validation datasets. A robust CADx algorithm should also involve global trainable data to minimise the introduction of bias. It is for these reasons that this is a planned international multicentre study.

The Investigators aim to develop a novel AI five class pathology prediction risk prediction tool that provides reliable information to identify cancer risk independent of the endoscopists skill.

These 5 categories are chosen because treatment options differ according to the polyp type and future check colonoscopy guidelines require these categories

DETAILED DESCRIPTION:
The use of artificial intelligence in computer-assisted detection (CADe) to detect polyps (pre-cancerous growths) during colonoscopy is gaining increasing interest and acceptance with multiple devices already in the mainstream market. The Investigator know already from work in other countries that detecting more polyps results in a reduced risk of bowel cancer for the patient having the procedure, in the years following their colonoscopy (ie. pre-cancerous growths were detected and removed). This has formed the basis of national bowel cancer screening programmes. With increased detection of colorectal polyps, there is a growing need to correctly identify the nature of the polyp to inform the risk of colorectal cancer with the polyp detected and also the potential future risk to the patient. Accurate polyp diagnosis is also required to determine the correct mode or removal-whether this does require removal at all (leading to conservation of costs and resources in a challenging current climate), whether endoscopic removal is possible and if so by what procedure, whether surgery is required.

Published data demonstrates that approximately one quarter of surgically removed colorectal polyps with patients undergoing major surgery were benign and therefore major surgery could have been avoided with these polyps removed endoscopically reducing the risk of complication and organ preservation for the patient.

Current polyp diagnosis techniques involve the use and interpretation of specialist dyes and magnification endoscopes which come with gaining expertise expertise with an associated learning curve and increased procedure time. It is for these reasons that despite being introduced in clinical practice, uptake of such techniques is limited and current methods of polyp risk stratification during colonoscopy without AI is suboptimal.

Current polyp diagnosis AI (CADx) algorithms are limited to smaller classification Current CADx platforms differentiate between cancerous and non-cancerous polyps which is of limited value in providing a personalised patient risk for colorectal cancer. The development of a multiclass algorithm is of greater complexity than a binary classification and requires larger training and validation datasets. A robust CADx algorithm should also involve global trainable data to minimise the introduction of bias. It is for these reasons that this is a planned international multicentre study

Prospective collection of data:

This study will be conducted alongside usual patient care, but will require research staff to enter data onto a secure web-based report form (REDCAP database). This means that participants will undergo exactly the same procedure, with no differences and no extra visits or data, than would have otherwise have occurred. Participants will be those patients that have been scheduled to have a colonoscopy for the standard reasons. Patients will be invited in the usual way for colonoscopy.

They may - where possible - be sent the PIS with their appointment letter (up to 6 weeks in advance). On arrival in the endoscopy unit, they will be approached by a member of the research team and given a copy of the PIS to read - up to an hour before their procedure. They will be provided face-to-face information and explanation, prior to written consent to allow their data to be collected in the database. As the study does not require any change or additional procedures, The investigator feel that an initial approach on arrival into the endoscopy unit will provide sufficient, appropriate time to consent, even if the PIS has not been read in advance (although it will be sent if possible). The only additional consideration will be the consent to recording of the video (no patient identifiable data will be transferred as part of this aspect).

Once the colonoscopy has been completed, there will be no additional visits.

ELIGIBILITY:
Inclusion Criteria:

- Above 18 years at inclusion Symptomatic or screening colonoscopy

Exclusion Criteria:

* Unable to provide informed consent.
* Colitis Associated Dysplasia
* Polyps at surgical anastomosis sites
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult (over 18 years) presenting for screening or symptomatic colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To achieve an overall accuracy of 85% for the five-classification lesion prediction algorithm. | 24 months
  Sensitivity and Specificity
Positive and negative predicted value | 24 months
  Assess the accuracy to the trained device

SECONDARY OUTCOMES:
Interobserver agreement of the endoscopists' prediction of histology of polyps during the annotation process. | 36 months
  We will analyse the calculate the histology agreement between the advance endoscopist
Sub-analysis of the polyp characteristics focused on different gender and ethnicity. | 36 months
  To assess if the prediction of patient gender, ethnicity, and age is possible with use of the developed CADx model.
This will be a sub analysis of an AI algorithm that is trained to predict polyp histology using the prospective data cohort. | 36 months
  A qualitative analysis of CADx incorrect diagnoses will also be conducted by a multidisciplinary panel to evaluate potential impact
Learned effects of AI augmented endoscopy on endoscopist optical diagnosis | 36 months
  We will evaluate if the use of AI during colonoscopy can be a learning tools for endoscopist

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided